CLINICAL TRIAL: NCT01348100
Title: An Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Two Iloperidone Depot Formulations Followed by a Dose-ranging Phase of One Selected Formulation in Schizophrenic Patients Given Depot Injections Every 28 Days
Brief Title: Safety, Tolerability, and Pharmacokinetics of Iloperidone Depot in Schizophrenic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CILO522E2101
Record Dates: First submitted 2011-04-28; First posted 2011-05-05 (Estimated); Results first posted 2013-10-08 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Iloperidone; Depot; Injection
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

ARMS (7):
- Iloperidone 50 mg crystalline formulation - Phase A (Experimental): Participants received a crystalline formulation of iloperidone 50 mg in a depot intramuscular (IM) injection 1 time. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 7 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone crystalline formulation; Drug: Oral iloperidone
- Iloperidone 125 mg crystalline formulation - Phase A (Experimental): Participants received a crystalline formulation of iloperidone 125 mg in a depot IM injection 1 time. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 7 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone crystalline formulation; Drug: Oral iloperidone
- Iloperidone 250 mg crystalline formulation - Phase B (Experimental): Participants received a crystalline formulation of iloperidone 250 mg in a depot IM injection 1 time. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 10 to 14 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone crystalline formulation; Drug: Oral iloperidone
- Iloperidone 250 mg microparticle formulation - Phase B (Experimental): Participants received a microparticle formulation of iloperidone 250 mg in a depot IM injection 1 time. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 10 to 14 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone microparticle formulation; Drug: Oral iloperidone
- Iloperidone 250 mg microparticle formulation - Phase C (Experimental): Participants received a microparticle formulation of iloperidone 250 mg in a depot IM injection 2 times 28 days apart. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 10 to 14 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone microparticle formulation; Drug: Oral iloperidone
- Iloperidone 500 mg microparticle formulation - Phase C (Experimental): Participants received a microparticle formulation of iloperidone 500 mg in a depot IM injection 2 times 28 days apart. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 10 to 14 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone microparticle formulation; Drug: Oral iloperidone
- Iloperidone 625 mg microparticle formulation - Phase C (Experimental): Participants received a microparticle formulation of iloperidone 625 mg in a depot IM injection 2 times 28 days apart. Prior to receiving IM iloperidone, participants were gradually titrated up with oral iloperidone for at least 10 to 14 days to stable doses of 12 to 24 mg daily.
  Interventions: Drug: Iloperidone microparticle formulation; Drug: Oral iloperidone

INTERVENTIONS:
Drug: Iloperidone crystalline formulation — Iloperidone was formulated as 100 µm crystals for IM depot injection.
  Arms: Iloperidone 125 mg crystalline formulation - Phase A; Iloperidone 250 mg crystalline formulation - Phase B; Iloperidone 50 mg crystalline formulation - Phase A
Drug: Iloperidone microparticle formulation — Iloperidone was formulated as microparticles for IM depot injection.
  Arms: Iloperidone 250 mg microparticle formulation - Phase B; Iloperidone 250 mg microparticle formulation - Phase C; Iloperidone 500 mg microparticle formulation - Phase C; Iloperidone 625 mg microparticle formulation - Phase C
Drug: Oral iloperidone — Prior to receiving an intramuscular (IM) injection of iloperidone, patients were gradually titrated up with oral iloperidone to stable doses of 12 to 24 mg daily. In Phase A, oral iloperidone dosing lasted for at least 7 days and, in Phases B and C, for at least 10 to 14 days.

SUMMARY:
This study is designed as a 3-part trial to evaluate the safety of a novel depot formulation of iloperidone, compare 2 depot dosage forms, and perform dose ranging of 1 chosen form in support of a monthly depot dosing regimen. In Phase A, the study is designed to evaluate the safety of a crystalline iloperidone depot formulation. In Phase B, the pharmacokinetic and safety profile of 2 depot clinical dosage forms will be compared, and 1 form will be selected for assessment in Phase C. Phase C of this study is designed to define the dose-exposure relationship of the selected form and to provide information that will permit a comparison of the risk-benefit ratio of several doses of the study drug to enable optimal dose selection for later studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia that have been stable for 3 months.

Exclusion Criteria:

* Women who can become or are currently pregnant or lactating.
* Hypersensitivity to iloperidone or related drugs.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iloperidone 50 mg Crystalline Formulation - Phase A | Iloperidone 125 mg Crystalline Formulation - Phase A | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C
Started | 2 | 2 | 15 | 15 | 15 | 16 | 16
Completed | 2 | 2 | 13 | 14 | 14 | 14 | 13
Not Completed | 0 | 0 | 2 | 1 | 1 | 2 | 3
Not completed — Subject Withdrew Consent | 0 | 0 | 2 | 0 | 1 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Effect | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Administrative Problems | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloperidone 50 mg Crystalline Formulation - Phase A | Iloperidone 125 mg Crystalline Formulation - Phase A | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C | Total
Number analyzed (Participants) | 2 | 2 | 15 | 15 | 15 | 16 | 16 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (2.83) | 35.5 (12.02) | 45.5 (14.81) | 43.5 (13.02) | 42.3 (10.62) | 41.3 (10.03) | 45.1 (11.21) | 43.3 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 5 | 4 | 6 | 5 | 3 | 25
  Male | 2 | 0 | 10 | 11 | 9 | 11 | 13 | 56

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Iloperidone Divided by the Average Plasma Concentration (Cav) of Iloperidone (Cmax/Cav) - Phase B
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. PK parameters were calculated from plasma concentration-time data using non-compartmental methods.
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: Ratio of Cmax to Cav
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
Ratio of Cmax to Cav | 1.91 (0.513) | 1.87 (0.554)

2. Primary Outcome: The Average Plasma Concentration (Cav) of Iloperidone - Phase C
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. Blood samples were collected after each depot injection. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Cav was calculated as AUC0-672h/672 h.
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C
Number analyzed (Participants) | 15 | 14 | 14
ng/mL
  Dose 1 - n = 15, 13, 12 | 3.73 (1.16) | 7.93 (5.29) | 11.8 (8.10)
  Dose 2 - n = 14, 14, 13 | 4.52 (1.50) | 10.1 (5.46) | 16.0 (7.12)

3. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Iloperidone - Phase B
Description: as for outcome 1
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hours
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
hours | 48.1 [0 to 169] | 168 [6 to 434]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Iloperidone - Phase B
Description: as for outcome 1
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
ng/mL | 6.25 (2.98) | 8.40 (3.49)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the End of the Dosing Period (AUCtau) of Iloperidone - Phase B
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. The area under the curve was calculated using a linear trapezoidal method. The end of the dosing period was 672 hours (28 days).
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
ng*h/mL | 2310 (1170) | 3190 (1670)

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Last Measurable Concentration (AUClast) of Iloperidone - Phase B
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. The area under the curve was calculated using a linear trapezoidal method.
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
ng*h/mL | 2890 (1380) | 3730 (1730)

7. Secondary Outcome: The Average Plasma Concentration (Cav) of Iloperidone - Phase B
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Cav was calculated as AUC0-672h/672 h.
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
ng/mL | 3.44 (1.74) | 4.74 (2.49)

8. Secondary Outcome: Duration That the Concentration of Iloperidone Was Above 4 ng/mL (Teff) - Phase B
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. The duration that the concentration of iloperidone was above 4 ng/mL was calculated by linear interpolation. PK/pharmacodynamic analysis performed in other studies suggests that iloperidone plasma levels of 4 ng/mL or above provide clinical efficacy.
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hours
Arm/Group | Iloperidone 250 mg Crystalline Formulation - Phase B | Iloperidone 250 mg Microparticle Formulation - Phase B
Number analyzed (Participants) | 13 | 14
hours | 150 [0 to 714] | 365 [0 to 801]

9. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Iloperidone - Phase C
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. Blood samples were collected after each depot injection. PK parameters were calculated from plasma concentration-time data using non-compartmental methods.
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hours
Arm/Group | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C
Number analyzed (Participants) | 15 | 14 | 14
hours
  Dose 1 - n = 15, 14, 14 | 48 [3 to 506] | 227 [3 to 601] | 192 [24 to 672]
  Dose 2 - n = 14, 14, 13 | 48 [24 to 266] | 207 [36 to 600] | 195 [48 to 385]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Iloperidone - Phase C
Description: as for outcome 9
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C
Number analyzed (Participants) | 15 | 14 | 14
ng/mL
  Dose 1 - n = 15, 14, 14 | 6.45 (2.29) | 15.2 (13.9) | 19.7 (15.8)
  Dose 2 - n = 14, 14, 13 | 8.15 (2.98) | 21.6 (19.6) | 29.2 (16.4)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the End of the Dosing Period (AUCtau) of Iloperidone - Phase C
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn pre-dose and at 3, 6, and 12 hours on Day 1; at 0 and 12 hours on Day 2; and on Days 3, 4, 6, 8, 10, 14, 18, 22, and 26 following administration of iloperidone. Blood samples were collected after each depot injection. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. The area under the curve was calculated using a linear trapezoidal method. The end of the dosing period was 672 hours (28 days).
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C
Number analyzed (Participants) | 15 | 14 | 14
ng*h/mL
  Dose 1 - n = 15, 13, 12 | 2500 (780) | 5330 (3560) | 7930 (5440)
  Dose 2 - n = 14, 14, 13 | 3040 (1010) | 6820 (3670) | 10700 (4790)

12. Secondary Outcome: The Average Plasma Concentration (Cav) of Iloperidone Divided by Dose - Phase C
Description: as for outcome 2
Time Frame: Pre-dose to 26 days post-dose
Population: Pharmacokinetic population: All participants with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Iloperidone 250 mg Microparticle Formulation - Phase C | Iloperidone 500 mg Microparticle Formulation - Phase C | Iloperidone 625 mg Microparticle Formulation - Phase C
Number analyzed (Participants) | 15 | 14 | 14
ng/mL/mg
  Dose 1 - n = 15, 13, 12 | 0.0156 (0.00464) | 0.0172 (0.0107) | 0.0196 (0.0125)
  Dose 2 - n = 14, 14, 13 | 0.0300 (0.0235) | 0.0242 (0.0129) | 0.0328 (0.0141)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline to the end of the study.
Description: Safety population: All participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment. One participant each in the Iloperidone 500 mg Microparticle Formulation - Phase C and the Iloperidone 625 mg Microparticle Formulation - Phase C groups did not receive iloperidone.
Groups:
- Iloperidone 50 mg Crystalline Formulation - Phase A Oral; Iloperidone 125 mg Crystalline Formulation - Phase A Oral: Prior to receiving an intramuscular (IM) injection of iloperidone, patients were gradually titrated up with oral iloperidone for at least 7 days to stable doses of 12 to 24 mg daily.
- Iloperidone 50 mg Crystalline Formulation - Phase A Depot: Participants received a crystalline formulation of iloperidone 50 mg in a depot intramuscular (IM) injection 1 time.
- Iloperidone 125 mg Crystalline Formulation - Phase A Depot: Participants received a crystalline formulation of iloperidone 125 mg in a depot IM injection 1 time.
- Iloperidone 250 mg Crystalline Formulation - Phase B Oral; Iloperidone 250 mg Microparticle Formulation - Phase B Oral; Iloperidone 250 mg Microparticle Formulation - Phase C Oral; Iloperidone 500 mg Microparticle Formulation - Phase C Oral; Iloperidone 625 mg Microparticle Formulation - Phase C Oral: Prior to receiving an intramuscular (IM) injection of iloperidone, patients were gradually titrated up with oral iloperidone for at least 10 to 14 days to stable doses of 12 to 24 mg daily.
- Iloperidone 250 mg Crystalline Formulation - Phase B Depot: Participants received a crystalline formulation of iloperidone 250 mg in a depot IM injection 1 time.
- Iloperidone 250 mg Microparticle Formulation - Phase B Depot: Participants received a microparticle formulation of iloperidone 250 mg in a depot IM injection 1 time.
- Iloperidone 250 mg Microparticle Formulation - Phase C Depot: Participants received a microparticle formulation of iloperidone 250 mg in a depot IM injection 2 times 28 days apart.
- Iloperidone 500 mg Microparticle Formulation - Phase C Depot: Participants received a microparticle formulation of iloperidone 500 mg in a depot IM injection 2 times 28 days apart.
- Iloperidone 625 mg Microparticle Formulation - Phase C Depot: Participants received a microparticle formulation of iloperidone 625 mg in a depot IM injection 2 times 28 days apart.
Arm/Group | Iloperidone 50 mg Crystalline Formulation - Phase A Oral | Iloperidone 125 mg Crystalline Formulation - Phase A Oral | Iloperidone 50 mg Crystalline Formulation - Phase A Depot | Iloperidone 125 mg Crystalline Formulation - Phase A Depot | Iloperidone 250 mg Crystalline Formulation - Phase B Oral | Iloperidone 250 mg Microparticle Formulation - Phase B Oral | Iloperidone 250 mg Crystalline Formulation - Phase B Depot | Iloperidone 250 mg Microparticle Formulation - Phase B Depot | Iloperidone 250 mg Microparticle Formulation - Phase C Oral | Iloperidone 500 mg Microparticle Formulation - Phase C Oral | Iloperidone 625 mg Microparticle Formulation - Phase C Oral | Iloperidone 250 mg Microparticle Formulation - Phase C Depot | Iloperidone 500 mg Microparticle Formulation - Phase C Depot | Iloperidone 625 mg Microparticle Formulation - Phase C Depot
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/15 | 0/15 | 2/14 | 1/14 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 1/2 | 2/2 | 9/15 | 10/15 | 4/14 | 8/14 | 11/15 | 9/15 | 9/15 | 13/15 | 12/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone 50 mg Crystalline Formulation - Phase A Oral (N=2) | Iloperidone 125 mg Crystalline Formulation - Phase A Oral (N=2) | Iloperidone 50 mg Crystalline Formulation - Phase A Depot (N=2) | Iloperidone 125 mg Crystalline Formulation - Phase A Depot (N=2) | Iloperidone 250 mg Crystalline Formulation - Phase B Oral (N=15) | Iloperidone 250 mg Microparticle Formulation - Phase B Oral (N=15) | Iloperidone 250 mg Crystalline Formulation - Phase B Depot (N=14) | Iloperidone 250 mg Microparticle Formulation - Phase B Depot (N=14) | Iloperidone 250 mg Microparticle Formulation - Phase C Oral (N=15) | Iloperidone 500 mg Microparticle Formulation - Phase C Oral (N=15) | Iloperidone 625 mg Microparticle Formulation - Phase C Oral (N=15) | Iloperidone 250 mg Microparticle Formulation - Phase C Depot (N=15) | Iloperidone 500 mg Microparticle Formulation - Phase C Depot (N=15) | Iloperidone 625 mg Microparticle Formulation - Phase C Depot (N=15)
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Social stay hospitalisation (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone 50 mg Crystalline Formulation - Phase A Oral (N=2) | Iloperidone 125 mg Crystalline Formulation - Phase A Oral (N=2) | Iloperidone 50 mg Crystalline Formulation - Phase A Depot (N=2) | Iloperidone 125 mg Crystalline Formulation - Phase A Depot (N=2) | Iloperidone 250 mg Crystalline Formulation - Phase B Oral (N=15) | Iloperidone 250 mg Microparticle Formulation - Phase B Oral (N=15) | Iloperidone 250 mg Crystalline Formulation - Phase B Depot (N=14) | Iloperidone 250 mg Microparticle Formulation - Phase B Depot (N=14) | Iloperidone 250 mg Microparticle Formulation - Phase C Oral (N=15) | Iloperidone 500 mg Microparticle Formulation - Phase C Oral (N=15) | Iloperidone 625 mg Microparticle Formulation - Phase C Oral (N=15) | Iloperidone 250 mg Microparticle Formulation - Phase C Depot (N=15) | Iloperidone 500 mg Microparticle Formulation - Phase C Depot (N=15) | Iloperidone 625 mg Microparticle Formulation - Phase C Depot (N=15)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection site exfoliation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 9
Injection site joint pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 8 | 9 | 10
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 5 | 1 | 2 | 4 | 1 | 3 | 4 | 1 | 2
Oromandibular dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Dissociation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obsessive thoughts (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Azoospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Ejaculation failure (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Painful ejaculation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retrograde ejaculation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 5 | 3 | 4 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone lesion excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.